CLINICAL TRIAL: NCT05597228
Title: Adapting and Testing an eHealth Platform to Deliver a Group Intervention for Young Adult Cancer Survivors
Brief Title: Tech-TYA: eHealth Platform to Deliver Group Intervention for YA Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000717
Record Dates: First submitted 2022-09-21; First posted 2022-10-28 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Cancer
Keywords: Neoplasms; Quality of life; Young adults
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral: Cognitive-Behavioral Stress Management and Health Education (Experimental): Weekly video conference groups led by a trained facilitator
  Interventions: Behavioral: Cognitive-Behavioral Stress Management and Health Education

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Stress Management and Health Education — Participants will attend group sessions with a trained facilitator held over videoconference. Sessions will each last 2 hours and be held once weekly for 10 weeks. Sessions will include Cognitive-Behavioral Stress Management and health education content.

SUMMARY:
The purpose of this study is to adapt a web-based platform to deliver a group intervention for young adult cancer survivors.

DETAILED DESCRIPTION:
In the first part of this study, the investigators adapted a website to deliver an evidence-based intervention for improving HRQOL for young adult cancer survivors, and then conducted usability testing sessions with young adult cancer survivors to get feedback on the website. In the second part of the study, the investigators will conduct a single-arm pilot trial in which the website will be used to deliver the intervention via weekly group meetings with a trained facilitator over the course of 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-39 years at the time of participation
2. Diagnosed with a primary cancer between 18-39 years old
3. Finished cancer treatment with curative intent 1 month to 5 years prior to enrollment (except hormone therapy)
4. NED and no anticipated/scheduled anti-cancer treatments at the time of enrollment (except hormone therapy)
5. Able to speak and read English
6. Able and willing to give informed consent
7. Access to internet or cellular connectivity with sufficient bandwidth to participate in videoconferences (Part 2 only)

Exclusion Criteria:

1. Ongoing or future anti-cancer treatments (beyond hormone therapy) are scheduled or anticipated
2. Documented or observable psychiatric or neurological disorders that could interfere with study participation (e.g., psychosis, active substance abuse)

Vulnerable populations will not be included in this study.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the eHealth intervention delivery | At the end of the 10-week intervention, overall and weekly satisfaction scores will be compiled
  Immediately after the intervention and each week participants will report their satisfaction with the full program through a brief survey.
Acceptability of the eHealth intervention delivery | At the end of the 10-week intervention
  Immediately after the intervention participants will report their satisfaction with the full program through a brief survey.
Acceptability of the eHealth intervention delivery | At the end of the 10-week intervention, the number of sessions attended will be recorded
  The number of sessions attended, out of a maximum of 10, will be recorded

SECONDARY OUTCOMES:
Change in health-related quality of life (HRQOL) from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the 27-item Functional Assessment of Cancer Therapy - General. Scores range from 0 to 108, with higher scores reflecting better quality of life.
Change in anxiety symptoms from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the Patient-Reported Outcomes Measurement Information System (PROMIS) Emotion Distress-Anxiety Short Form 4a. Raw scores are converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate more symptoms of anxiety.
Change in perceived cognitive function from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the PROMIS Cognitive Function Short Form 4a. Raw scores are converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate better perceived cognitive function.
Change in depression symptoms from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the PROMIS Cognitive Function Short Form 4a. Raw scores are converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate better perceived cognitive function.
Change in perceived emotional support from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the PROMIS Emotional Support Short Form 4a. Raw scores are converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate greater perceived emotional support.
Change in fatigue from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the PROMIS Fatigue Short Form 4a. Raw scores are converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate more fatigue.
Change in pain interference from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the PROMIS Pain Interference Short Form 4a. Raw scores are converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate more pain interference.
Change in patient-reported physical function from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the PROMIS Physical Function Short Form 4a. Raw scores are converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate better patient-reported physical function.
Change in pain intensity from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the PROMIS Pain Intensity 1a. Scores range from 0 to 10, with higher scores indicating greater pain intensity.
Change in cancer-related distress from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the 22-item Impact of Event Scale-Revised. Scores range from 0 to 88, with higher scores indicating greater cancer-related distress.
Change in stress management self-efficacy skills from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete subscales from the Measure of Current Status. Subscale scores range from 0 to 8, 0 to 12, or 0 to 20 depending on the subscale. Higher scores indicate more of the construct being assessed.
Change in coping from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the Brief Coping Orientation to Problems Experienced scale, which yields 14 two-item subscales. Subscale scores range from 2 to 8, with higher scores indicating greater usage of the coping strategy being assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fox RS, Badger TA, Moya S, Gudenkauf LM, Nelson MA, O'Neill RM, Leete JJ, Friedman SE, Katsanis E, Victorson DE, Sanford SD, Penedo FJ, Antoni MH, Oswald LB. An HRQOL Proof-Of-Concept Analysis of the eHealth TOGETHER Intervention for Adolescent and Young Adult Cancer Survivors: A Brief Report. Psychooncology. 2025 Jul;34(7):e70234. doi: 10.1002/pon.70234. PMID 40879639
- [Derived] Fox RS, Torres TK, Badger TA, Katsanis E, Yang D, Sanford SD, Victorson DE, Yanez B, Penedo FJ, Antoni MH, Oswald LB. Delivering a Group-Based Quality of Life Intervention to Young Adult Cancer Survivors via a Web Platform: Feasibility Trial. JMIR Cancer. 2024 Dec 4;10:e58014. doi: 10.2196/58014. PMID 39631050